CLINICAL TRIAL: NCT02424903
Title: European Prosthetic Joint Infection Cohort Study (EPJIC): Evaluation of the Treatment Approach for Hip, Knee and Shoulder Prosthetic Joint Revision Surgery
Brief Title: European Prosthetic Joint Infection Cohort Study- Hip, Knee and Shoulder Prosthetic Joint Infection
Acronym: EPJIC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pro-Implant Foundation (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: PJI04/2014
Record Dates: First submitted 2015-03-24; First posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Prosthesis-related Infections
Keywords: infection; prosthesis; hip; knee; shoulder
MeSH Terms: conditions — Prosthesis-Related Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with prosthetic joint infection: Patients admitted for a septic revision surgery
- without prosthetic joint infection: Patients admitted for an aseptic revision surgery

SUMMARY:
The purpose of the study is to compare different approaches for the treatment of prosthetic joint revisions and to optimize the outcomes in patients with prosthetic joint infections (PJI) by improving the treatment concept of PJI.

DETAILED DESCRIPTION:
The aim of the study is to assess the impact of different surgical and antibiotic therapies on patients admitted for a septic or aseptic revision of the hip, knee or shoulder prosthesis. The decision whether the implant will be retained or removed or antimicrobial treatment is based on criteria of each participating center specialists.The success of different treatment algorithms will be measured in terms of infection free interval, functional outcome and quality of life. All consecutive patients who need a revision surgery to the hip, knee or shoulder will be included. Furthermore the study will investigate different diagnostic tests (microbiological and histological) for the diagnosis and the discrimination of septic and aseptic causes in prosthesis failures. Pathogens (microorganisms isolated from puncture of the joint, tissue samples sonication fluid and blood) will be collected to establish a biobank.The samples are obtained preoperatively and intraoperatively as part of routine care practice. The study is not randomized.

ELIGIBILITY:
Inclusion Criteria:

* subject is older than 18 years of Age
* written informed consent has been obtained
* subject Needs a Revision surgery of the hip, knee or shoulder prosthesis

Exclusion Criteria:

* subject is currently enrolled in another investigational study
* inability to read and understand the participant's Information
* subject is younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to hospital
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Infection outcome | 12 months after surgery
  The infection-free status is defined as absence of clinical (e.g. no fistula), laboratory (e.g. normal C-reactive protein) and radiological signs of infection (e.g. no septic loosening).

SECONDARY OUTCOMES:
Functional outcome | 12 months after surgery
  by HARRIS HIP SCORE, CONSTANT SHOULDER SCORE, KNEE SOCIETY SCORE, OXFORD HIP SCORE, OXFORD KNEE SCORE, QUICK DASH SCORE
lifequality evaluation | 12 months after surgery
  by EQ5D5l-score

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Trampuz, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité, Berlin, Berlin, Germany